CLINICAL TRIAL: NCT00175279
Title: A Cluster Randomized Trial to Assess the Impact of Opinion Leader Endorsed Evidence Summaries on Improving Quality of Prescribing for Patients With Chronic Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Heritage Foundation for Medical Research (Other); Institute of Health Economics, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISRCTN26365328; IHE#102
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Coronary Disease; Ischemic Heart Disease; Heart Failure
Keywords: coronary disease; heart failure; quality improvement; knowledge translation; opinion leaders
MeSH Terms: conditions — Coronary Disease; Myocardial Ischemia; Heart Failure

INTERVENTIONS:
Behavioral: Opinion leader generated and endorsed evidence summaries

SUMMARY:
BACKGROUND: Although much has been written about the influence of local opinion leaders on clinical practice, there have been few controlled studies of their effect, and almost none have attempted to change prescribing in the community for chronic conditions such as congestive heart failure (CHF) or ischemic heart disease (IHD). These two conditions are common and there is very good evidence about how to best prevent morbidity and mortality - and very good evidence that quality of care is, in general, suboptimal. Practice audits have demonstrated that about half of eligible CHF patients are prescribed ACE inhibitors (and fewer still reaching appropriate target doses) and less than one-third of patients with established IHD are prescribed statins (with many fewer reaching recommended cholesterol targets). It is apparent that interventions to improve quality of prescribing are urgently needed.

HYPOTHESIS: An intervention that consists of patient-specific one-page evidence summaries, generated and then endorsed by local opinion leaders, will be able to change prescribing practices of community-based primary care physicians.

DESIGN: A single centre randomized controlled trial comparing an opinion leader intervention to usual care. Based on random allocation of all physicians in one large Canadian health region, patients with CHF or IHD (not receiving ACE inhibitors or statins, respectively) recruited from community pharmacies will be allocated to intervention or usual care. The primary outcome is improvement in prescription of proven efficacious therapies for CHF (ACE inhibitors) or IHD (statins) within 6 months of the intervention.

DETAILED DESCRIPTION:
BACKGROUND: Although much has been written about the influence of local opinion leaders on clinical practice, there have been few controlled studies of their effect, and almost none have attempted to change prescribing in the community for chronic conditions such as congestive heart failure (CHF) or ischemic heart disease (IHD). These two conditions are common and there is very good evidence about how to best prevent morbidity and mortality - and very good evidence that quality of care is, in general, suboptimal. Practice audits have demonstrated that about half of eligible CHF patients are prescribed ACE inhibitors (and fewer still reaching appropriate target doses) and less than one-third of patients with established IHD are prescribed statins (with many fewer reaching recommended cholesterol targets). It is apparent that interventions to improve quality of prescribing are urgently needed.

HYPOTHESIS: An intervention that consists of patient-specific one-page evidence summaries, generated and then endorsed by local opinion leaders, will be able to change prescribing practices of community-based primary care physicians.

DESIGN: A single centre randomized controlled trial comparing an opinion leader intervention to usual care. Based on random allocation of all physicians in one large Canadian health region, patients with CHF or IHD (not receiving ACE inhibitors or statins, respectively) recruited from community pharmacies will be allocated to intervention or usual care. The primary outcome is improvement in prescription of proven efficacious therapies for CHF (ACE inhibitors) or IHD (statins) within 6 months of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HF or IHD who are not currently taking the study medications of interest (ACE inhibitors/angiotensin receptor blockers for HF or statins for IHD) and whose primary care physicians are part of the study population

Exclusion Criteria:

* Patients who are unable or unwilling to give informed consent,
* previously taken the study medications according to dispensing records
* allergy or intolerance to study medications
* residents of long-term care facilities
* unable to confirm a diagnosis of either HF or IHD
* primary care physician has already contributed 5 patients to the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2002-01; Study Completion 2005-04

PRIMARY OUTCOMES:
The primary outcome measure will be the "improvement" of prescribing for efficacious therapies in patients with a chronic cardiovascular disease within six months of the intervention.

SECONDARY OUTCOMES:
1. Condition-specific "improvement" in prescribing after 6 months.
2. "Optimization" of dosage for each of the medications prescribed (i.e., ACE inhibitors or angiotensin receptor blockers and statins).
3. Patient adherence
4. Subgroup analyses based on condition, age, and sex.

CONTACTS AND LOCATIONS:
Overall Officials: Sumit R Majumdar, MD, MPH, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Majumdar SR, McAlister FA, Tsuyuki RT. A cluster randomized trial to assess the impact of opinion leader endorsed evidence summaries on improving quality of prescribing for patients with chronic cardiovascular disease: rationale and design [ISRCTN26365328]. BMC Cardiovasc Disord. 2005 Jun 27;5(1):17. doi: 10.1186/1471-2261-5-17. PMID 15982421
- [Result] Majumdar SR, Tsuyuki RT, McAlister FA. Impact of opinion leader-endorsed evidence summaries on the quality of prescribing for patients with cardiovascular disease: a randomized controlled trial. Am Heart J. 2007 Jan;153(1):22.e1-8. doi: 10.1016/j.ahj.2006.07.030. PMID 17174632